CLINICAL TRIAL: NCT02776137
Title: Postoperative Concurrent Chemoradiotherapy With Docetaxel for High-Risk Squamous Cell Carcinoma of Head and Neck，A Non-Randomized Phase II Trial
Brief Title: Postoperative Concurrent Chemoradiotherapy With Docetaxel for High-Risk Squamous Cell Carcinoma of Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016HNRT001
Record Dates: First submitted 2016-05-11; First posted 2016-05-18 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Head-and-neck Cancer; Squamous Cell Carcinoma
Keywords: Docetaxel; Concurrent Chemoradiotherapy; High-Risk; Squamous Cell Carcinoma; Head-and-Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Docetaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel Group (Experimental): Concurrent Chemoradiotherapy With Docetaxel
  Interventions: Drug: Docetaxel; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Docetaxel — Docetaxel: 20mg/m2/w for 6 weeks
Radiation: Intensity-modulated radiotherapy — a total dose of 60Gy in 30 fractions over 6 weeks
  Other Names: IMRT

SUMMARY:
This is a non-randomized, phase II, open label study of postoperative concurrent chemoradiotherapy with docetaxel for high-risk squamous cell carcinoma of the head and neck(HNSCC).The primary purpose of this study is to evaluate the efficacy and safety of concurrent chemoradiotherapy with docetaxel in HNSCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the head and neck.Site of tumor origin in the oral cavity, oropharynx, larynx, or hypopharynx (excluding nasopharynx, or sinuses)
2. Gross total resection, with pathology demonstrating one or more of the following risk factors:

   1. Histologic extracapsular nodal extension
   2. Histologic involvement of ≥ 2 regional lymph nodes
   3. Invasive cancer seen on microscopic evaluation of the resection margin, with no evidence of gross tumor residual
3. No evidence of distant metastases
4. No synchronous or concurrent head and neck primary tumors
5. Karnofsky score over 60
6. Adequate organ function including the following:

   1. Absolute neutrophil count (ANC) >= 1.5 * 10^9/l
   2. Platelets count >= 100 * 10^9/l
   3. Hemoglobin >= 10 g/dl
   4. AST and ALT <= 2.5 times institutional upper limit of normal (ULN)
   5. Total bilirubin <= 1.5 times institutional ULN
   6. Creatinine clearance >= 50 ml/min
   7. Serum creatine <= 1 times ULN
7. Signed written informed consent

Exclusion Criteria:

1. Evidence of distant metastasis
2. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
3. Other previous cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
4. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
5. Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 2 years

SECONDARY OUTCOMES:
overall survival rate | 2 years
  from date of enrollment until date of first death from any cause, assessed up to 2 years
Acute toxicity profiles, graded according to the NCI CTCAE version 3.0 | up to 6-7 weeks
  Number of participants with treatment-related acute toxicity as assessed weekly by CTCAE v3.0 during the course of treatment
Late toxicity profiles, graded according to the NCI CTCAE version 3.0 | up to 2 years
  Number of participants with treatment-related late toxicity as assessed every 3 months by CTCAE v3.0 up to 2 years
Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Core 35 (EORTC QLQ-HN35) during the concurrent treatment | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  QoL score will be documented on each weekend during the course of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Zhu, M.D., Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li R, Jiang W, Dou S, Zhong L, Sun J, Zhang C, Zhu G. A Phase 2 Trial of Chemoradiation Therapy Using Weekly Docetaxel for High-Risk Postoperative Oral Squamous Cell Carcinoma Patients. Int J Radiat Oncol Biol Phys. 2020 Jul 1;107(3):462-468. doi: 10.1016/j.ijrobp.2020.02.464. Epub 2020 Feb 29. PMID 32126267